CLINICAL TRIAL: NCT01734772
Title: Investigation of Drug-drug Interaction of Dabigatran and Ticagrelor Under Steady State Conditions in Healthy Male Subjects
Brief Title: Investigation of Drug-drug Interaction of Dabigatran and Ticagrelor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.142; 2012-002656-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Ticagrelor

ARMS (3):
- Reference (Part 1/A, Part 2/C) (Experimental): multiple doses of dabigatran (alone)
  Interventions: Drug: dabigatran etexilate
- Test 1 (Part 1/Treatment B) (Experimental): concomitant administration of dabigatran and ticagrelor
  Interventions: Drug: dabigatran etexilate; Drug: ticagrelor
- Test 2 (Part 2/Treatment D) (Experimental): staggered administration of ticagrelor and dabigatran
  Interventions: Drug: ticagrelor; Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — multiple doses of dabigatran
  Arms: Test 1 (Part 1/Treatment B)
Drug: dabigatran etexilate — medium dose dabigatran
  Arms: Reference (Part 1/A, Part 2/C)
Drug: ticagrelor — loading dose of ticagrelor
  Arms: Test 1 (Part 1/Treatment B)
Drug: ticagrelor — multiple doses of ticagrelor
  Arms: Test 1 (Part 1/Treatment B)
Drug: ticagrelor — loading dose of ticagrelor
  Arms: Test 2 (Part 2/Treatment D)
Drug: dabigatran etexilate — single dose of dabigatran
  Arms: Test 2 (Part 2/Treatment D)

SUMMARY:
To investigate the pharmacokinetic and pharmacodynamic interaction of dabigatran and ticagrelor under steady state conditions; to investigate the effect of staggered administration of ticagrelor loading dose on dabigatran exposure (in Part II)

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects.

Exclusion criteria:

1. Any relevant deviation from healthy conditions.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.142.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: In part 1, 110 mg dabigatran etexilate were dosed twice daily to steady state and a dabigatran PK profile was taken on day 3 (reference). On the day after the reference treatment, ticagrelor treatment was added starting with the concomitant administration of a 180 mg ticagrelor loading dose followed by 90 mg ticagrelor twice daily. Dabigatran PK profiles were taken on day 1 of the test treatment and day 4 of the test treatment.
- Part 2: In part 2, 110 mg dabigatran etexilate were dosed twice daily to steady state and a dabigatran PK profile was taken on day 3 (reference). On the day after the reference treatment, 180 mg ticagrelor were given 2 hours after the morning dose of 110 mg dabigatran etexilate and dabigatran PK profile were taken on this day 1 of the test treatment.
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 24 | 24
Completed | 23 | 21
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set which includes all subjects who were documented to have received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.2) | 28.6 (7.1) | 28.3 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Total Dabigatran: Area Under the Concentration-time Curve at Steady State Over the Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of dabigatran etexilate in plasma at steady state over the uniform dosing interval τ (AUCτ,ss).
Time Frame: 47.55, 48.30,49, 49.30,50,50.30,51,52,54,56, 60 hours
Population: Pharmacokinetic set: This subject set included all subjects in the TS who provided at least 1 observation for at least 1 PK endpoint without important protocol violations relevant to the evaluation of bioavailability and who had not vomiting at or before 2 times the median tmax,ss of the trial medications on PK study days of both trial parts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Dabigratan Etexilate 110mg Bid Alone - Part 1; Dabigratan Etexilate 110mg Bid Alone - Part 2: Dabigatran Etexilate 110mg twice daily (bid) for 3 days
- Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1: Single loading dose of Ticagrelor 180 mg on day 1 together with Dabigatran Etexilate 110mg bid.
- Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1: Multiple dosing of 90 mg bid on days 2 and 3 and 90mg on day 4 together with Dabigatran Etexilate 110mg bid on days 2 and 3 and 110mg in the morning on day 4.
- Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2: Dabigatran Etexilate 110mg morning dose followed by 180mg Ticagrelor 2 hours later.
Arm/Group | Dabigratan Etexilate 110mg Bid Alone - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1 | Dabigratan Etexilate 110mg Bid Alone - Part 2 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2
Number analyzed (Participants) | 24 | 23 | 23 | 23 | 21
ng*h/mL | 551 (59.0) | 817 (43.3) | 689 (55.1) | 660 (39.6) | 844 (43.4)
Statistical Analysis 1: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 1 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.9456, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; geometric Mean Ratio = 149.38, 90% CI [124.388 to 179.383], Standard Deviation 37.6 — The dispersion value is actually the intraindividual gCV
Statistical Analysis 2: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 1 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.5481, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; geometric Mean Ratio = 126.47, 90% CI [107.363 to 148.967], Standard Deviation 33.3 — The dispersion value is actually the intraindividual gCV
Statistical Analysis 3: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 2 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.5665, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; geometric Mean Ratio = 127.01, 90% CI [108.047 to 149.295], Standard Deviation 31.6 — The dispersion value is actually the intraindividual gCV

2. Primary Outcome: Total Dabigatran: Maximum Measured Concentration at Steady State (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss).
Time Frame: 47.55, 48.30,49, 49.30,50,50.30,51,52,54,56, 60 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigratan Etexilate 110mg Bid Alone - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1 | Dabigratan Etexilate 110mg Bid Alone - Part 2 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2
Number analyzed (Participants) | 24 | 23 | 23 | 23 | 21
ng/mL | 83.6 (69.3) | 136 (45.4) | 106 (65.1) | 97.6 (46.5) | 121 (45.2)
Statistical Analysis 1: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 1 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.9841, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; geometric Mean Ratio = 164.74, 90% CI [133.945 to 202.619], Standard Deviation 42.9 — The dispersion value is actually the intraindividual gCV
Statistical Analysis 2: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 1 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.6003, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; geometric Mean Ratio = 128.61, 90% CI [106.370 to 155.495], Standard Deviation 39.0 — The dispersion value is actually the intraindividual gCV
Statistical Analysis 3: Comparison: Dabigratan Etexilate 110mg Bid Alone - Part 2 vs Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.4656, ANOVA — p-value for ratio outside interval 80% - 125%; Adjustment for effects 'subject' and 'treatment'; gMean Ratio = 123.82, 90% CI [102.695 to 149.288], Standard Deviation 36.9 — The dispersion value is actually the intraindividual gCV

ADVERSE EVENTS:
Time Frame: 11 days
Groups:
- Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1: Multiple dosing of 90 mg bid on days 2 and 3 and 90mg on day 4 together with Dabigatran Etexilate 110mg bid on days 2 and 3 and 110mg once on day 4.
Arm/Group | Dabigratan Etexilate 110mg Bid Alone - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1 | Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1 | Dabigratan Etexilate 110mg Bid Alone - Part 2 | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23 | 2/24 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigratan Etexilate 110mg Bid Alone - Part 1 (N=24) | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 1 (N=23) | Dabigatran Etexilate 110mg Bid + Ticagrelor 90mg Bid - Part 1 (N=23) | Dabigratan Etexilate 110mg Bid Alone - Part 2 (N=24) | Dabigatran Etexilate 110mg Bid + Ticagrelor 180 mg - Part 2 (N=21)
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.